CLINICAL TRIAL: NCT03127644
Title: A Phase 2/3 Multicenter, Dose-response Study to Assess Efficacy and Safety of ZS (Sodium Zirconium Cyclosilicate), in Japanese Patients With Hyperkalemia
Brief Title: ZS Ph2/3 Dose-response Study in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9482C00002
Record Dates: First submitted 2017-04-05; First posted 2017-04-25 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-02

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium Zirconium Cyclosilicate (ZS) 5g (Experimental): Suspension administered 5g orally three times daily for 48 hours.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS) 5g
- Sodium Zirconium Cyclosilicate (ZS) 10g (Experimental): Suspension administered 10g orally three times daily for 48 hours.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS) 10g
- Placebo (Placebo Comparator): Placebo suspension administered orally placebo three times daily for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (ZS) 5g — Suspension administered 5g orally three times daily for 48 hours.
  Arms: Sodium Zirconium Cyclosilicate (ZS) 5g
Drug: Sodium Zirconium Cyclosilicate (ZS) 10g — Suspension administered 10g orally three times daily for 48 hours.
  Arms: Sodium Zirconium Cyclosilicate (ZS) 10g
Drug: Placebo — Placebo suspension administered orally placebo three times daily for 48 hours.
  Arms: Placebo

SUMMARY:
To assess efficacy of 5 g three times daily (TID) and 10 g TID ZS versus placebo in Japanese patients with hyperkalemia (serum potassium [S-K] ≥ 5.1 mmol/L and ≤ 6.5 mmol/L).

DETAILED DESCRIPTION:
Patients not receiving any therapy for hyperkalemia and with 2 consecutive i-STAT potassium values of ≥ 5.1 mmol/L and ≤ 6.5 mmol/L will be enrolled and randomized 1:1:1 to receive ZS 5 g, ZS 10 g, or placebo TID for 48 hours.

Throughout the study most potassium values will be measured at fasting before taking study drug. Nothing should be taken by mouth except water, coffee or tea, with or without milk and/or sugar, and essential medications, prior to the blood collection for a minimum of 8 hours. Potassium level should be determined by both i-STAT and the Central Laboratory on all occasions. Treatment decisions (eg, stopping rules) will be made based on i-STAT potassium values, as these provide clinical sites with a real-time measurement. Statistical analyses on the study data will in principle be based on S-K values as measured by the central laboratory.

Safety and tolerability will be assessed on an ongoing basis. Standard study assessments including blood potassium, clinical chemistry (including calcium, magnesium, sodium, phosphate, creatinine, bicarbonate, and blood urea nitrogen [BUN]) and hematology parameters, urinalysis, vital signs, physical examinations, and electrocardiograms (ECGs) will be assessed during the study at the time points specified in the assessments schedule. All women of childbearing potential will have a urine pregnancy test prior to enrollment and at their End of Study (EOS) visit.

Stopping rules will be implemented to ensure subjects discontinue the study treatment and receive alternative therapy in case of significant hyperkalemia, hypokalemia, or significant cardiac arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Patients aged ≥18. For patients aged <20 years, a written informed consent should be obtained from the patient and his or her legally acceptable representative.
* Two consecutive i-STAT potassium values, measured 60 (± 10) minutes apart, both values should be ≥ 5.1 mmol/L and ≤ 6.5 mmol/L and measured within 1 day before the first dose of study drug on Study Day 1.
* Ability to have repeated blood draws or effective venous catheterization.
* Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of ZS/matching placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Cause or symptoms of pseudohyperkalemia, such as

  1. hemolyzed blood specimen due to excessive fist clenching to make veins prominent
  2. hemolyzed blood specimen due to difficult or traumatic venepuncture
  3. history of severe leukocytosis or thrombocytosis
* Patients treated with lactulose, rifaximin, or other non-absorbed antibiotics for hyperammonemia within 7 days prior to first dose of study drug on Study Day 1
* Patients treated with resins (such as sevelamer hydrochloride, sodium polystyrene sulfonate [SPS; e.g. Kayexalate®] or calcium polystyrene sulfonate [CPS]), calcium acetate, calcium carbonate, or lanthanum carbonate, within 7 days prior to the first dose of study drug
* Patients with a life expectancy of less than 3 months
* Patients who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the patients' tasks associated with the protocol
* Female patients who are pregnant, lactating, or planning to become pregnant
* Patients who have an active or history of diabetic ketoacidosis
* Presence of any condition which, in the opinion of the investigator, places the patient at undue risk or potentially jeopardizes the quality of the data to be generated
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry
* Patients with cardiac arrhythmias that require immediate treatment
* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Japan (24):
  - Research Site, Chiba
  - Research Site, Hanyu-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Hitachi-Naka
  - Research Site, Ina-shi
  - Research Site, Kagoshima
  - Research Site, Kahoku-gun
  - Research Site, Kamakura-shi
  - Research Site, Kanazawa
  - Research Site, Kasugai-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Koga-shi
  - Research Site, Kusatsu-shi
  - Research Site, Matsudo-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Omura-shi
  - Research Site, Shimajiri-gun
  - Research Site, Shizuoka
  - Research Site, Yakushi
  - Research Site, Yotsukaido-shi

REFERENCES:
- [Derived] Kashihara N, Nishio T, Osonoi T, Saka Y, Imasawa T, Ohtake T, Mizuno H, Shibagaki Y, Kim H, Yajima T, Sarai N. Correction of serum potassium with sodium zirconium cyclosilicate in Japanese patients with hyperkalemia: a randomized, dose-response, phase 2/3 study. Clin Exp Nephrol. 2020 Dec;24(12):1144-1153. doi: 10.1007/s10157-020-01937-1. Epub 2020 Aug 10. PMID 32779057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients not receiving any therapy for hyperkalaemia and with 2 consecutive potassium values of ≥ 5.1 millimoles/litre (mmol/L) and ≤ 6.5 mmol/L (as measured by i-STAT, a portable blood analyser) were enrolled into 24 study sites in Japan from June 2017 to February 2018.
Pre-assignment Details: 103 patients were randomised 1:1:1 to receive double-blind treatment of sodium zirconium cyclosilicate (ZS) 5 grams (g) three times daily (TID), ZS 10 g TID, or placebo TID for 48 hours.
Groups:
- ZS 5 g TID: ZS suspension was administered 5 g orally TID for 48 hours.
- ZS 10 g TID: ZS suspension was administered 10 g orally TID for 48 hours.
- Placebo TID: Placebo suspension was administered orally TID for 48 hours.
Period: Overall Study
Arm/Group | ZS 5 g TID | ZS 10 g TID | Placebo TID
Started | 34 | 36 | 33
Completed | 34 | 36 | 31
Not Completed | 0 | 0 | 2
Not completed — Study-specific withdrawal criteria | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set included all patients randomised in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ZS 5 g TID | ZS 10 g TID | Placebo TID | Total
Number analyzed (Participants) | 34 | 36 | 33 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.4 (7.9) | 71.1 (7.6) | 76.1 (6.8) | 73.2 (7.7)
Age, Customized [Number; unit: Participants]
  <55 years | 0 | 1 | 0 | 1
  55 to 64 years | 7 | 4 | 1 | 12
  ≥65 years | 27 | 31 | 32 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 10 | 26
  Male | 26 | 28 | 23 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 36 | 33 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 34 | 36 | 33 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Exponential Rate of Change in Serum Potassium (S-K) Values During the Initial 48 Hours of Study Drug Treatment
Description: Blood samples for determination of potassium were collected pre-dose, and at 1, 2, and 4 hours post Dose 1 on Day 1. An additional sample was collected at 90 minutes post Dose 2 on Day 1 if i-STAT potassium values at the 4-hour post Dose 1 time point was ≥ 6.1 or <4.0 mmol/L. On Day 2 samples were analysed pre-dose, and 1 and 4 hours post Dose 1. S-K levels were analysed at the Central Laboratory.
  Natural logarithm of S-K from 0 to 48 hours post dose are modelled by the random coefficients model including fixed effects of intercept, time, time x treatment and patient-level random effects for time and intercept. Exponential rate of change refers to the slope estimate from the random coefficients model.
Time Frame: From 0 to 48 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Mean (Standard Error); unit: log (mmol/L) / hour
Arm/Group | ZS 5 g TID | ZS 10 g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
log (mmol/L) / hour | -0.00273 (0.000276) | -0.00508 (0.000269) | -0.00012 (0.000288)
Statistical Analysis 1: Comparison: ZS 10 g TID vs Placebo TID; Exponential rate of change in S-K through to 48 hours was analysed with a mixed effect model (random slope model); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Confirmatory testing proceeded sequentially (ZS 10g TID, then ZS 5g TID); Treatment difference in slopes = -0.00496, 95% CI 2-sided [-0.00571 to -0.00420], Standard Error of Mean 0.000380 — Negative exponential rate of change relative to placebo indicates more rapid reduction (correction) of S-K
Statistical Analysis 2: Comparison: ZS 5 g TID vs Placebo TID; Exponential rate of change in S-K through to 48 hours was analysed with a mixed effect model (random slope model); Test type: Superiority; p < 0.001, Mixed Models Analysis; Confirmatory testing proceeded sequentially (ZS 10g TID, then ZS 5g TID); Treatment difference in slopes = -0.00261, 95% CI 2-sided [-0.00337 to -0.00185], Standard Error of Mean 0.000385 — Negative exponential rate of change relative to placebo indicates more rapid reduction (correction) of S-K

2. Secondary Outcome: Percentage of Patients Who Achieved Normokalaemia at 48 Hours
Description: The percentage of patients who achieved normokalaemia (normalisation of S-K values to between 3.5 mmol/L and 5.0 mmol/L, inclusive) at 48 hours after start of dosing was determined. Patients with missing S-K values at 48 hours were regarded as not normokalaemic.
Time Frame: At 48 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Number; unit: Percentage of Patients
Groups:
- ZS 10g TID: ZS suspension was administered 10 g orally TID for 48 hours.
Arm/Group | ZS 5 g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Percentage of Patients | 85.3 | 91.7 | 15.2
Statistical Analysis 1: Comparison: ZS 5 g TID vs Placebo TID; Logistic regression model including treatment and baseline S-K as explanatory variables was used; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 46.495, 95% CI 2-sided [10.142 to 213.152]
Statistical Analysis 2: Comparison: ZS 10g TID vs Placebo TID; Logistic regression model including treatment and baseline S-K as explanatory variables was used; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 71.835, 95% CI 2-sided [13.497 to 382.337]

3. Secondary Outcome: Exponential Rate of Change in S-K Values During the Initial 24 Hours of Study Drug Treatment
Description: Blood samples for determination of potassium were collected pre-dose, and at 1, 2, and 4 hours post Dose 1 on Day 1. An additional sample was collected at 90 minutes post Dose 2 on Day 1 if i-STAT potassium values at the 4-hour post Dose 1 time point was ≥ 6.1 or <4.0 mmol/L. On Day 2 samples were analysed pre-dose, and 1 and 4 hours post Dose 1. S-K levels were analysed at the Central Laboratory. Natural logarithm of S-K from 0 to 24 hours post dose are modelled by the random coefficients model including fixed effects of intercept, time, time x treatment and patient-level random effects for time and intercept. Exponential rate of change refers to the slope estimate from the random coefficients model.
Time Frame: From 0 to 24 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Mean (Standard Error); unit: log (mmol/L) / hour
Arm/Group | ZS 5 g TID | ZS 10 g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
log (mmol/L) / hour | -0.00234 (0.000468) | -0.00403 (0.000457) | -0.00002 (0.000489)
Statistical Analysis 1: Comparison: ZS 5 g TID vs Placebo TID; Exponential rate of change in S-K through to 24 hours was analysed with a mixed effect model (random slope model); Test type: Superiority; p = 0.0004, Mixed Models Analysis; Treatment difference in slopes = -0.00231, 95% CI 2-sided [-0.00359 to -0.00104], Standard Error of Mean 0.000645 — Negative exponential rate of change relative to placebo indicates more rapid reduction (correction) of S-K
Statistical Analysis 2: Comparison: ZS 10 g TID vs Placebo TID; Exponential rate of change in S-K through to 24 hours was analysed with a mixed effect model (random slope model); Test type: Other; p < 0.0001, Mixed Models Analysis; Treatment difference in slopes = -0.00401, 95% CI 2-sided [-0.00527 to -0.00275], Standard Error of Mean 0.000637 — Negative exponential rate of change relative to placebo indicates more rapid reduction (correction) of S-K

4. Secondary Outcome: Percentage of Patients Who Achieved Normokalaemia at 24 Hours
Description: The percentage of patients who achieved normokalaemia (normalisation of S-K values to between 3.5 mmol/L and 5.0 mmol/L, inclusive) at 24 hours after start of dosing was determined. Patients with missing S-K values at 24 hours were regarded as not normokalaemic.
Time Frame: At 24 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Number; unit: Percentage of Patients
Arm/Group | ZS 5 g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Percentage of Patients | 35.3 | 83.3 | 27.3
Statistical Analysis 1: Comparison: ZS 5 g TID vs Placebo TID; Logistic regression model including treatment and baseline S-K as explanatory variables was used; Test type: Superiority; p = 0.6167, Regression, Logistic; Odds Ratio (OR) = 1.347, 95% CI 2-sided [0.419 to 4.329]
Statistical Analysis 2: Comparison: ZS 10g TID vs Placebo TID; Logistic regression model including treatment and baseline S-K as explanatory variables was used; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 15.334, 95% CI 2-sided [4.006 to 58.697]

5. Secondary Outcome: Percentage of Patients Who Achieved Normokalaemia at Each Scheduled Potassium Assessment Time Point
Description: The percentage of patients who achieved normokalaemia (normalisation of S-K values to between 3.5 mmol/L and 5.0 mmol/L, inclusive) at each each scheduled potassium assessment time point after the start of dosing was determined. Patients with missing S-K values were regarded as not normokalaemic.
Time Frame: From baseline to end of study (9 days).
Population: The full analysis set included all patients randomised in the study.
Measure: Number; unit: Percentage of Patients
Arm/Group | ZS 5 g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Percentage of Patients
  Baseline | 2.9 | 5.6 | 0.0
  1 hour after first dose | 29.4 | 47.2 | 21.2
  2 hours after first dose | 41.2 | 58.3 | 42.4
  4 hours after first dose | 44.1 | 63.9 | 42.4
  24 hours after first dose | 35.3 | 83.3 | 27.3
  25 hours after first dose | 73.5 | 97.2 | 18.2
  28 hours after first dose | 67.6 | 97.2 | 36.4
  48 hours after first dose | 85.3 | 91.7 | 15.2
  End of study (Last dose + 7 days) | 55.9 | 61.1 | 27.3

6. Secondary Outcome: Mean Change From Baseline in S-K Values at All Measured Time Intervals
Description: Blood samples for determination of potassium were collected pre-dose, and at 1, 2, and 4 hours post Dose 1 on Day 1. An additional sample was collected at 90 minutes post Dose 2 on Day 1 if i-STAT potassium values at the 4-hour post Dose 1 time point was ≥ 6.1 or <4.0 mmol/L. On Day 2 samples were analysed pre-dose, and 1 and 4 hours post Dose 1. S-K levels were analysed locally using i-STAT devices, and at the Central Laboratory. S-K values measured at each time point and end of study visit were recorded and mean change from baseline is displayed.
Time Frame: From baseline to end of study (9 days).
Population: The full analysis set included all patients randomised in the study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ZS 5 g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
mmol/L
  1 hour after first dose | -0.20 (0.34) | -0.37 (0.35) | -0.13 (0.32)
  2 hours after first dose: number analyzed (Participants) | 34 | 36 | 32
  2 hours after first dose | -0.41 (0.28) | -0.50 (0.40) | -0.33 (0.30)
  4 hours after first dose: number analyzed (Participants) | 34 | 36 | 32
  4 hours after first dose | -0.40 (0.32) | -0.53 (0.36) | -0.43 (0.31)
  24 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  24 hours after first dose | -0.51 (0.30) | -0.69 (0.38) | -0.22 (0.35)
  25 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  25 hours after first dose | -0.74 (0.31) | -1.00 (0.45) | -0.27 (0.31)
  28 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  28 hours after first dose | -0.72 (0.35) | -1.12 (0.39) | -0.41 (0.43)
  48 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  48 hours after first dose | -0.83 (0.31) | -1.30 (0.48) | -0.24 (0.34)
  End of study (Last dose + 7 days) | -0.56 (0.38) | -0.66 (0.52) | -0.20 (0.59)

7. Secondary Outcome: Mean Percent Change From Baseline in S-K Values at All Measured Time Intervals
Description: Blood samples for determination of potassium were collected pre-dose, and at 1, 2, and 4 hours post Dose 1 on Day 1. An additional sample was collected at 90 minutes post Dose 2 on Day 1 if i-STAT potassium values at the 4-hour post Dose 1 time point was ≥ 6.1 or <4.0 mmol/L. On Day 2 samples were analysed pre-dose, and 1 and 4 hours post Dose 1. S-K levels were analysed locally using i-STAT devices, and at the Central Laboratory. S-K values measured at each time point and end of study visit were recorded and mean percent change from baseline is displayed.
Time Frame: From baseline to end of study (9 days).
Population: The full analysis set included all patients randomised in the study.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ZS 5 g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Percent change
  1 hour after first dose | -3.61 (6.28) | -6.72 (6.29) | -2.32 (5.60)
  2 hours after first dose: number analyzed (Participants) | 34 | 36 | 32
  2 hours after first dose | -7.46 (5.04) | -9.07 (6.88) | -6.06 (5.40)
  4 hours after first dose: number analyzed (Participants) | 34 | 36 | 32
  4 hours after first dose | -7.08 (5.65) | -9.70 (6.53) | -7.77 (5.62)
  24 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  24 hours after first dose | -8.98 (5.33) | -12.51 (6.30) | -3.81 (6.24)
  25 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  25 hours after first dose | -13.20 (5.42) | -18.06 (7.05) | -4.77 (5.66)
  28 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  28 hours after first dose | -12.90 (6.10) | -20.47 (6.38) | -7.21 (7.61)
  48 hours after first dose: number analyzed (Participants) | 34 | 36 | 31
  48 hours after first dose | -14.81 (5.08) | -23.64 (8.27) | -4.06 (5.93)
  End of study (Last dose + 7 days) | -9.85 (6.51) | -11.89 (9.07) | -3.15 (9.99)

8. Secondary Outcome: Time to Normalisation in S-K Values
Description: The distribution of time to normalisation of S-K values (defined as S-K values between 3.5 mmol/L and 5.0 mmol/L, inclusive) was measured. A patient who reached at least one S-K within normal range was counted as an event regardless of S-K value after that time point. Patients who did not achieve normokalaemia within 48 hours were censored.
Time Frame: From 0 to 48 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- ZS 5g TID: ZS suspension was administered 5 g orally TID for 48 hours.
Arm/Group | ZS 5g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Hours | 3.883 [1.767 to 23.083] | 1.758 [1.000 to 3.967] | 3.867 [1.917 to NA] — Upper limit not reached.
Statistical Analysis 1: Comparison: ZS 5g TID vs Placebo TID; Test type: Superiority; p = 0.0586, Log Rank — Nominal p value
Statistical Analysis 2: Comparison: ZS 10g TID vs Placebo TID; Test type: Superiority; p = 0.0006, Log Rank — Nominal p value

9. Secondary Outcome: Time to a Decrease in S-K Levels of 0.5 mmol/L
Description: The median time (hours) for S-K values to decrease by 0.5 mmol/L was measured.
Time Frame: From 0 to 48 hours.
Population: The full analysis set included all patients randomised in the study.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | ZS 5g TID | ZS 10g TID | Placebo TID
Number analyzed (Participants) | 34 | 36 | 33
Hours | 3.883 [1.933 to 19.767] | 2.892 [1.083 to 4.100] | 4.050 [1.983 to 23.667]
Statistical Analysis 1: Comparison: ZS 5g TID vs Placebo TID; Test type: Superiority; p = 0.0250, Log Rank — Nominal p value
Statistical Analysis 2: Comparison: ZS 10g TID vs Placebo TID; Test type: Superiority; p = 0.0064, Log Rank — Nominal p value

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were reported from Day 1 to Day 3 inclusive.
Arm/Group | ZS 5 g TID | ZS 10 g TID | Placebo TID
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 4/34 | 5/36 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZS 5 g TID (N=34) | ZS 10 g TID (N=36) | Placebo TID (N=33)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (5) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03127644/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03127644/SAP_001.pdf